CLINICAL TRIAL: NCT05825287
Title: The Effect of Patient Education Given by Teach-Back Method on Managing Chemotherapy Symptoms and Quality of Life-Randomized Controlled Study
Brief Title: The Effect of Patient Education Given by Teach-Back Method on Managing Chemotherapy Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, BELKIS GULLU GUCUYENER, Principal investigator, Marmara University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Marmara U
Record Dates: First submitted 2023-03-30; First posted 2023-04-24 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Teach-Back Communication
Keywords: Teach-Back; Life quality; chemotherapy side effects
MeSH Terms: conditions — Teach-Back Communication | interventions — Anger Management Therapy

STUDY DESIGN:
Intervention Model Description: The model of research is quantitative. Participants are experimental because they are randomly selected to the interference and control group. It is a randomized controlled clinical study, a group of interventions and controls, to determine the impact of the first-time education in patients who have been diagnosed with cancer and have been treated for chemotherapy to manage symptoms and determine the quality of life of patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trained by teaching back method (Active Comparator): The course method will determine which group to assign the first patient to meet the criteria for inclusion in the study by the researcher. Subsequent patients will be distributed to groups in turn. It is planned to include 40 participants in the study, as losses may occur among the participants. The study will begin on the day that cancer-treated participants receive chemotherapy for the first time. Considering that the participants would be more comfortable and the training would be healthy, the training was planned 30 minutes before the application. The training was planned by the researcher in the chemotherapy case manager's room as face-to-face meetings with each participant separately. Each training will be accompanied by a chemotherapy case manager. Training time is between 20-30 minutes as planned.
  Interventions: Other: Trained by teaching back method
- Management training (Experimental): The course method will determine which group to assign the first patient to meet the criteria for inclusion in the study by the researcher. Subsequent patients will be distributed to groups in turn. It is planned to include 40 participants in the study, as losses may occur among the participants. The study will begin on the day that cancer-treated participants receive chemotherapy for the first time. Considering that the participants would be more comfortable and the training would be healthy, the training was planned 30 minutes before the application. The training was planned by the researcher in the chemotherapy case manager's room as face-to-face meetings with each participant separately. Each training will be accompanied by a chemotherapy case manager. Training time is between 20-30 minutes as planned.
  Interventions: Other: Management training

INTERVENTIONS:
Other: Trained by teaching back method — in chemotherapy symptom management training, 2 groups will be created and a group will be given normal symptom management training, and the other group will be trained by teaching back method to assess the symptom control and quality of life after the chemotherapy training that patients have received and evaluate the effect of the teaching back method
  Arms: Trained by teaching back method
Other: Management training — Management training
  Arms: Management training

SUMMARY:
.The aim of this study is to evaluate the effectiveness of the education method given by using the documents shaped by the teach-back method in the management of the frequently encountered side effects in chemotherapy treatment and to develop an effective method that health professionals can use in patient education.

DETAILED DESCRIPTION:
Cancer is one of the most common groups of diseases in the world today that human beings have to deal with. The lack of exact treatment, as well as the presence of a wide range of cancer types, makes treatment algorithms difficult and prolonging treatment processes. The prime treatment options for the treatment currently used are surgical treatment, radiotherapy and chemotherapy. Although surgical treatment is on the forefront of early cancer patients, radiation therapy and chemotherapy treatments are currently making progress and progress. The variety of medications used, the use of drugs with different actuators, and even the combination of different methods such as radiotherapy and chemotherapy in therapy, can increase the chances of success, but can lead to serious side effects. This reduces patient compliance and may lead to the end of treatments. Research of the methods and behaviors to improve patient/patient relatives' compliance and participation in treatment has gained speed, and studies have become widespread, noting the importance of these models, although studies for finding groups of low-side effects drugs are still in progress. When it comes to treatment and patient care, the center of the circle is the nurses who are the primary care giver. The most important task is for nurses to continue the treatment process effectively and to eliminate compliance problems for patient/patient relatives. The correct approaches to managing the treatment of a disease group with increased side-effect insidance such as cancer will increase the quality of life and treatment adaptation process of patients, allowing the treatment to end as soon as possible. Particularly during chemotherapy treatment, nausea, vomiting, indigestion, abdominal pain, fatigue, etc. in the management of complaints such as, it should be the main task of nurses working in the field to describe problems and methods of dealing with patients/patients before treatment. Brochure for treatment and possible side effects in the majority of treatment centers, etc. there are documents, but often documented by medical terminology, these documents lead to confusion in the patient/patient vicinity and are unable to serve their intended use. Most of the time, it is thought that the patient and his relatives have been trained and learned. But what he learned from education is not questioned. The aim of this study is to evaluate the effectiveness of the training method provided using the documentation shaped by the way that you describe what is common to the management of side effects in chemotherapy treatment and to develop an effective method that health care personnel can use in patient education.

ELIGIBILITY:
Inclusion Criteria:

* First time chemotherapy,
* Patients over 18 years old
* Patients agree to participate in research
* Knowing and understanding Turkish
* IV and oral chemotherapy treatment
* Lack of communication problems and cognitive deficiency

Exclusion Criteria:

* He has been treated for chemotherapy before
* To receive radiation therapy with chemotherapy treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Edmonton Symptom Diagnosis Scale will be used to determine the effect of patient education given by the teack-back method on the management of symptoms between successive chemotherapy sessions. | Average 1 year
  In the Edmonton Symptom Diagnostic Scale, various symptoms such as pain, fatigue, nausea, sadness, anxiety, insomnia, loss of appetite, feeling well, shortness of breath, changes in the skin and nails, wounds in the mouth, numbness in the hands and other problems are questioned. The person completing the scale evaluates his/her own situation with a score between 0 and 10. 0 denotes the best case, 10 denotes the worst case.
The EQ-5D Quality of life scale will be used to determine the effect of patient education given by the teack-back method on the quality of life between consecutive chemotherapy sessions. | Average 1 year
  The EQ-5D is a self-report scale developed by the EuroQoL group, the Western European quality of life research community. It consists of two parts. Chapter 1 defines the health profile in 5 dimensions. (mobility, self-care, usual daily activities, pain/discomfort, and anxiety/depression) Each dimension includes 3 statements according to difficulty level. (1 some problem, 2 moderate, 3 a lot of problems) Section 2 includes the visual analog scale (VAS), in which respondents rate their current health status on a scale of 0 to 100. It is easy to apply and is completed in a short time.

CONTACTS AND LOCATIONS:
Overall Officials: Bilgi GULSEVEN KARABACAK, doctors, Principal Investigator — Marmara University
Locations (1):
- Ozel Anadolu Sağlik Merkezi, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I will not present individual participant data to other researchers.

REFERENCES:
- [Background] Yen PH, Leasure AR. Use and Effectiveness of the Teach-Back Method in Patient Education and Health Outcomes. Fed Pract. 2019 Jun;36(6):284-289. PMID 31258322
- See also: The Agency for Healthcare Research and Quality's (AHRQ) core competencies are Data and Analytics, Health Systems Research, and Practice Improvement. — http://www.ahrq.gov